CLINICAL TRIAL: NCT01006304
Title: A Double-blind, Randomized, Placebo-controlled, Crossover Study to Evaluate the Effects of JNJ-39439335 (a TRPV1 Antagonist) in Healthy Male Adult Subjects on the Paradoxical Pain Induced by a Thermal Grill
Brief Title: An Exploratory Study to Assess the Effects of JNJ-39439335 on the Relief of Pain Using a Thermal-Grill Experimental Model
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Clinical Leader
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: CR016666
Record Dates: First submitted 2009-10-29; First posted 2009-11-02 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2010-07

CONDITIONS: Pain
Keywords: JNJ-39439335; Placebo; Pain; Pain Measurements; Adults; Men
MeSH Terms: conditions — Pain; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: JNJ-39439335, Placebo

SUMMARY:
This exploratory study will use a thermal-grill experimental model to assess the effects of JNJ-39439335 (50 mg, single oral dose) on the relief of pain.

DETAILED DESCRIPTION:
This exploratory study will use a thermal-grill experimental model to assess the effects of JNJ-39439335 (50 mg, single oral dose) on the relief of pain. The study drug will be tested in healthy adult males to find out if a single 50 mg oral dose of JNJ-39439335 will be better than placebo (an inactive substance, like a sugar pill) in relieving pain. Study volunteers will experience the pain sensation (the illusion of pain) as a result of placing the palm of the hand on a small device that consists of harmless warm and cool flat metal bars known as a thermal grill. Volunteers will receive JNJ-39439335 or its matching placebo in the study unit on Day 1 of each of the 2 treatment periods. The treatment sequence for each volunteer will be assigned randomly (like flipping a coin). On the dosing day, the pain sensation will be induced and the following outcome measures will be assessed before dosing and at 4 hours after dosing: (1) volunteer's heat pain threshold [HPT] and cold pain threshold [CPT], i.e., the hot or the cold temperature at which it begins to elicit pain, (2) the intensity and the unpleasantness of the pain sensation resulting from simultaneous application of a warm temperature [4 C below HPT] and a cold temperature [4 C above CPT], (3) the intensity of non-painful warm and cold sensations following application of temperatures 4 C below HPT or 4 C above CPT, respectively, and (4) the intensity of pain following application of temperatures 2 C above HPT and 2 C below CPT. All of these assessments will be performed at a constant room temperature of approximately 21 C. During the trial volunteers will be closely monitored for safety, including the evaluation of adverse events, vital signs, 12-lead ECG, clinical laboratory testing (hematology and serum chemistry), and full neurological examination. Two blood samples for the measurement of JNJ-39439335 plasma concentrations will be collected immediately before and immediately after the thermal-grill assessments. At approximately 6 hours post-dose, volunteers will be discharged from the study unit. The study duration for each volunteer is approximately 9 weeks, including a screening phase that starts within 3 weeks before the first study drug administration, a washout of at least 3 weeks between the 2 treatment periods, and a final follow-up visit that will take place at approximately 3 weeks after the last study drug administration. Each volunteer will receive a single oral dose of JNJ-39439335 (50 mg) or placebo tablet on Day 1 of each of the 2 treatment periods. The study duration for each subject is ~9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy man with body-mass-index of 18.5 to 30 kg/m2, inclusive

Exclusion Criteria:

* Men who smoke or use tobacco within 3 months prior to the first study drug administration, and/or have a positive cotinine test result at Screening
* and men who are not considered healthy based on the ECG, vital signs, physical examinations, and laboratory tests.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-06; Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The effects of JNJ-39439335 on the relief of paradoxical pain (the illusion of pain) | at predose and at 4 hours postdose

SECONDARY OUTCOMES:
The effects of JNJ-39439335 on the non-painful cold and warm sensations corresponding respectively to the cold and warm temperatures used to induce paradoxical pain | at predose and at 4 hours postdose in each of the 2 treatment periods
The effects of JNJ-39439335 on the normal cold- and heat-pain induced by supra-threshold cold and heat stimuli. | at predose and at 4 hours postdose in each of the 2 treatment periods

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.